CLINICAL TRIAL: NCT00000625
Title: A Randomized, Double-Blind Phase II/III Trial of Monotherapy vs. Combination Therapy With Nucleoside Analogs in HIV-Infected Persons With CD4 Cells of 200-500/mm3
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Bristol-Myers Squibb (Industry); Glaxo Wellcome (Industry)
Responsible Party: Sponsor
Masking: Double | Purpose: Treatment
Other Study IDs: ACTG 175; 11150 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Zalcitabine; Didanosine; Drug Therapy, Combination; AIDS-Related Complex; Antiviral Agents; Zidovudine
MeSH Terms: conditions — HIV Infections; AIDS-Related Complex | interventions — Zidovudine; Zalcitabine; Didanosine

INTERVENTIONS:
Drug: Zidovudine
Drug: Zalcitabine
Drug: Didanosine

SUMMARY:
To determine the efficacy and safety of zidovudine ( AZT ) versus didanosine ( ddI ), AZT plus ddI, and AZT plus zalcitabine ( ddC ) in preventing disease progression in HIV-infected patients with CD4 counts of 200-500 cells/mm3.

DETAILED DESCRIPTION:
Patients are randomized to receive AZT alone, AZT and ddI, AZT and ddC, or ddI alone for at least 2 years. Patients who develop AIDS or whose CD4 count falls to 50 percent or less of baseline are crossed over to another treatment arm.

PER AMENDMENT 4/5/95: Study treatment will be available until 10/31/95 at the latest for patients still taking study medications on 4/30/95, so that follow-up trials may be completed and approved.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* PCP prophylaxis, M. tuberculosis prophylaxis, short courses of acyclovir, chronic suppressive acyclovir, pneumovax or Hib vaccine, antibiotics, rEPO and G-CSF for grade 3 or worse anemia and neutropenia, systemic corticosteroids for < 21 days, regularly prescribed medications, and vitamins or herbal therapies.

Patients must have:

* HIV infection without AIDS with CD4 200-500 cells/mm3.

PER AMENDMENT 4/5/95:

* Patients must have remained on ACTG 175 study treatment through 4/30/95 and meet toxicity management criteria for continuing treatment. Subjects taking ACTG 175 crossover treatment are eligible.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions are excluded:

* Current AIDS-related condition other than minimal KS, grade 2 or worse peripheral neuropathy, and malignancy requiring systemic therapy.

Concurrent Medication:

Excluded:

* Other anti-HIV drugs, biologic response modifiers other than rEPO and G-CSF, systemic cytotoxic chemotherapy, chronic systemic corticosteroids, or any drug that affects AZT glucuronidation or clearance.

Concurrent Treatment:

Excluded:

* Radiotherapy other than limited local therapy to skin.

Patients with the following prior conditions are excluded:

* AIDS-related condition other than minimal KS; intolerance to AZT, ddI, or ddC at study doses; and acute or chronic pancreatitis.

Prior Medication:

Excluded:

* Acute therapy for an infection or other medical illness within the past 14 days.

Current alcohol abuse.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2100
Dates: Study Completion 1995-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katzenstein D, Study Chair; Hammer S, Study Chair
Locations (58):
- United States (56):
  - Alabama Therapeutics CRS, Birmingham, Alabama
  - USC CRS, Los Angeles, California
  - UCLA CARE Center CRS, Los Angeles, California
  - Children's Hosp. & Research Ctr. Oakland, Ped. Clinical Research Ctr. & Research Lab., Oakland, California
  - Stanford CRS, Palo Alto, California
  - UCSD Maternal, Child, and Adolescent HIV CRS, San Diego, California
  - Ucsd, Avrc Crs, San Diego, California
  - Ucsf Aids Crs, San Francisco, California
  - Santa Clara Valley Med. Ctr., San Jose, California
  - San Mateo County AIDS Program, San Mateo, California
  - Harbor-UCLA Med. Ctr. CRS, Torrance, California
  - University of Colorado Hospital CRS, Aurora, Colorado
  - Howard University Hosp., Div. of Infectious Diseases, ACTU, Washington D.C., District of Columbia
  - Univ. of Miami AIDS CRS, Miami, Florida
  - Emory Univ. Hemophilia Program Office, Atlanta, Georgia
  - Univ. of Hawaii at Manoa, Leahi Hosp., Honolulu, Hawaii
  - Northwestern University CRS, Chicago, Illinois
  - Cook County Hosp. CORE Ctr., Chicago, Illinois
  - Rush Univ. Med. Ctr. ACTG CRS, Chicago, Illinois
  - Indiana Univ. School of Medicine, Infectious Disease Research Clinic, Indianapolis, Indiana
  - Methodist Hosp. of Indiana, Indianapolis, Indiana
  - Univ. of Iowa Healthcare, Div. of Infectious Diseases, Iowa City, Iowa
  - Tulane Hemophilia Treatment Ctr., New Orleans, Louisiana
  - Tulane Med. Ctr. - Charity Hosp. of New Orleans, ACTU, New Orleans, Louisiana
  - Tulane/LSU Maternal/Child CRS, New Orleans, Louisiana
  - Johns Hopkins Adult AIDS CRS, Baltimore, Maryland
  - Massachusetts General Hospital ACTG CRS, Boston, Massachusetts
  - Brigham and Women's Hosp., Div. of Infectious Disease, Boston, Massachusetts
  - HMS - Children's Hosp. Boston, Div. of Infectious Diseases, Boston, Massachusetts
  - Bmc Actg Crs, Boston, Massachusetts
  - Beth Israel Deaconess - East Campus A0102 CRS, Boston, Massachusetts
  - Beth Israel Deaconess Med. Ctr., ACTG CRS, Boston, Massachusetts
  - Hennepin County Med. Ctr., Div. of Infectious Diseases, Minneapolis, Minnesota
  - University of Minnesota, ACTU, Minneapolis, Minnesota
  - St. Louis ConnectCare, Infectious Diseases Clinic, St Louis, Missouri
  - Washington U CRS, St Louis, Missouri
  - Univ. of Nebraska Med. Ctr., Durham Outpatient Ctr., Omaha, Nebraska
  - NJ Med. School CRS, Newark, New Jersey
  - SUNY - Buffalo, Erie County Medical Ctr., Buffalo, New York
  - Beth Israel Med. Ctr. (Mt. Sinai), New York, New York
  - NY Univ. HIV/AIDS CRS, New York, New York
  - Cornell University A2201, New York, New York
  - Memorial Sloan-Kettering Cancer Ctr., New York, New York
  - NYU Med. Ctr., Dept. of Medicine, New York, New York
  - Univ. of Rochester ACTG CRS, Rochester, New York
  - Unc Aids Crs, Chapel Hill, North Carolina
  - Carolinas HealthCare System, Carolinas Med. Ctr., Charlotte, North Carolina
  - Duke Univ. Med. Ctr. Adult CRS, Durham, North Carolina
  - Regional Center for Infectious Disease, Wendover Medical Center CRS, Greensboro, North Carolina
  - Wake County Health and Human Services CRS, Raleigh, North Carolina
  - Univ. of Cincinnati CRS, Cincinnati, Ohio
  - Case CRS, Cleveland, Ohio
  - MetroHealth CRS, Cleveland, Ohio
  - The Ohio State Univ. AIDS CRS, Columbus, Ohio
  - Hosp. of the Univ. of Pennsylvania CRS, Philadelphia, Pennsylvania
  - University of Washington AIDS CRS, Seattle, Washington
- Puerto Rico-AIDS CRS, San Juan, Puerto Rico
- Mbeya Med. Research Program, Mbeya Referral Hosp. CRS, Mbeya, Tanzania

REFERENCES:
- [Background] Havlir DV, Richman DD. Viral dynamics of HIV: implications for drug development and therapeutic strategies. Ann Intern Med. 1996 Jun 1;124(11):984-94. doi: 10.7326/0003-4819-124-11-199606010-00006. PMID 8624066
- [Background] Hammer SM, Katzenstein DA, Hughes MD, Gundacker H, Schooley RT, Haubrich RH, Henry WK, Lederman MM, Phair JP, Niu M, Hirsch MS, Merigan TC. A trial comparing nucleoside monotherapy with combination therapy in HIV-infected adults with CD4 cell counts from 200 to 500 per cubic millimeter. AIDS Clinical Trials Group Study 175 Study Team. N Engl J Med. 1996 Oct 10;335(15):1081-90. doi: 10.1056/NEJM199610103351501. PMID 8813038
- [Background] Simpson DM, Katzenstein DA, Hughes MD, Hammer SM, Williamson DL, Jiang Q, Pi JT. Neuromuscular function in HIV infection: analysis of a placebo-controlled combination antiretroviral trial. AIDS Clinical Group 175/801 Study Team. AIDS. 1998 Dec 24;12(18):2425-32. doi: 10.1097/00002030-199818000-00011. PMID 9875580
- [Background] Zidovudine, didanosine, and zalcitabine in the treatment of HIV infection: meta-analyses of the randomised evidence. HIV Trialists' Collaborative Group. Lancet. 1999 Jun 12;353(9169):2014-25. PMID 10376616
- [Background] Katzenstein DA, Hughes MD, Albrecht M, Liou SH, Murphy R, Balfour H, Para M, Hammer S; ACTG 302 Study Team. Virologic and CD4 cell response to zidovudine or zidovudine and lamivudine following didanosine treatment of human immunodeficiency virus infection. AIDS Res Hum Retroviruses. 2001 Feb 10;17(3):203-10. doi: 10.1089/088922201750063115. PMID 11177402
- [Background] Justice AC, Holmes W, Gifford AL, Rabeneck L, Zackin R, Sinclair G, Weissman S, Neidig J, Marcus C, Chesney M, Cohn SE, Wu AW; Adult AIDS Clinical Trials Unit Outcomes Committee. Development and validation of a self-completed HIV symptom index. J Clin Epidemiol. 2001 Dec;54 Suppl 1:S77-90. doi: 10.1016/s0895-4356(01)00449-8. PMID 11750213
- [Background] Katzenstein DA, Hammer SM, Hughes MD, Gundacker H, Jackson JB, Fiscus S, Rasheed S, Elbeik T, Reichman R, Japour A, Merigan TC, Hirsch MS. The relation of virologic and immunologic markers to clinical outcomes after nucleoside therapy in HIV-infected adults with 200 to 500 CD4 cells per cubic millimeter. AIDS Clinical Trials Group Study 175 Virology Study Team. N Engl J Med. 1996 Oct 10;335(15):1091-8. doi: 10.1056/NEJM199610103351502. PMID 8813039
- [Background] Fiscus SA, Hughes MD, Lathey JL, Pi T, Jackson B, Rasheed S, Elbeik T, Reichman R, Japour A, Byington R, Scott W, Griffith BP, Katzenstein DA, Hammer SM. Changes in virologic markers as predictors of CD4 cell decline and progression of disease in human immunodeficiency virus type 1-infected adults treated with nucleosides. AIDS Clinical Trials Group Protocol 175 Team. J Infect Dis. 1998 Mar;177(3):625-33. doi: 10.1086/514248. PMID 9498441
- [Background] Currier JS, Spino C, Grimes J, Wofsy CB, Katzenstein DA, Hughes MD, Hammer SM, Cotton DJ. Differences between women and men in adverse events and CD4+ responses to nucleoside analogue therapy for HIV infection. The Aids Clinical Trials Group 175 Team. J Acquir Immune Defic Syndr. 2000 Aug 1;24(4):316-24. doi: 10.1097/00126334-200008010-00003. PMID 11015147
- [Background] Kastrissios H, Suarez JR, Katzenstein D, Girard P, Sheiner LB, Blaschke TF. Characterizing patterns of drug-taking behavior with a multiple drug regimen in an AIDS clinical trial. AIDS. 1998 Dec 3;12(17):2295-303. doi: 10.1097/00002030-199817000-00011. PMID 9863872
- [Background] Lathey JL, Hughes MD, Fiscus SA, Pi T, Jackson JB, Rasheed S, Elbeik T, Reichman R, Japour A, D'Aquila RT, Scott W, Griffith BP, Hammer SM, Katzenstein DA. Variability and prognostic values of virologic and CD4 cell measures in human immunodeficiency virus type 1-infected patients with 200-500 CD4 cells/mm(3) (ACTG 175). AIDS Clinical Trials Group Protocol 175 Team. J Infect Dis. 1998 Mar;177(3):617-24. doi: 10.1086/514250. PMID 9498440